CLINICAL TRIAL: NCT06117033
Title: The Effect of Preoperative Routine Patient Education and Video-assisted Mobilization Training on Postoperative Mobillity, Anxiety Level and Pain in Patients Who Will Undergo Coronary Artery Bypass Graft Surgery
Brief Title: The Effect of Video-assisted Mobilisation Training on Mobility, Anxiety and Pain After Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Namik Kemal University (Other)
Responsible Party: Principal Investigator, Merve Tosun, Nurse, Namik Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MTosun
Record Dates: First submitted 2023-10-19; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Anxiety; Postoperative Pain
Keywords: coronary artery bypass graft; pain; mobility; anxiety
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Preoperative routine patient education and video-assisted mobilization training were given to patients undergoing coronary artery bypass graft surgery.
  Interventions: Other: video assisted mobilization training
- control group (No Intervention): Patients in the control group received only routine patient education.

INTERVENTIONS:
Other: video assisted mobilization training — Preoperative video-assisted mobilization training was given to patients undergoing coronary artery bypass graft surgery
  Arms: experimental group

SUMMARY:
This study is a Randomized Controlled trial.The aim of this study was to investigate the effect of preoperative routine patient education and video-assisted mobilization training on postoperative mobility, anxiety level and pain in patients undergoing coronary artery bypass graft surgery.

Hypotheses of the study:

H1= Routine patient education and video-assisted mobilization training have an effect on postoperative anxiety level in patients undergoing coronary artery bypass graft surgery.

H2= Routine patient education and video-assisted mobilization training have an effect on postoperative mobility in patients undergoing coronary artery bypass graft surgery.

H3= Routine patient education and video-assisted mobilization training have an effect on postoperative pain in patients undergoing coronary artery bypass graft surgery.

DETAILED DESCRIPTION:
This study is a Randomized Controlled trial. The study consists of 80 patients, 40 control and 40 study group. Patients in the experimental group who underwent coronary artery bypass graft surgery completed the "State Trait Anxiety Scale" in the preoperative period.

Then, video-assisted mobilization training was given together with routine patient training.After the patient underwent surgery, the "State Trait Anxiety Scale" was completed again before the first mobilization.After the first mobilization, "Patient Mobility Scale" and "Observer Mobility Scale" were completed."State Trait Anxiety Scale" was used again on the 2nd postoperative day before mobilization."Patient Mobility Scale" and "Observer Mobility Scale" were used after the patient was mobilized.

Patients in the control group who underwent coronary artery bypass graft surgery completed the "State Trait Anxiety Scale" in the preoperative period.Routine patient education was then given.After the patient underwent surgery, the "State Trait Anxiety Scale" was completed again before the first mobilization.After the first mobilization, "Patient Mobility Scale" and "Observer Mobility Scale" were completed. The "State Trait Anxiety Scale" was used again before mobilization on the 2nd postoperative day.After the patient was mobilized, "Patient Mobility Scale" and "Observer Mobility Scale" were used.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary artery bypass graft surgery,
* Patients aged 18 years and older,
* Patients who can speak Turkish,
* Patients without a diagnosis of cognitive and psychiatric disorders that prevent them from expressing themselves,
* Patients open to communication,
* Patients who volunteered to participate in the study and gave verbal and written informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
postoperative anxiety | up to six months
  The effects of routine patient education and video-assisted mobilization training on postoperative anxiety in patients undergoing coronary artery bypass graft surgery were investigated. State Trait Anxiety Scale was used to measure the level of postoperative anxiety. The scale consists of two parts: "State Anxiety Scale" and "Trait Anxiety Scale". The State Anxiety Scale consists of a total of 20 statements. It defines the state anxiety of the individual. The individual is asked to express how he/she feels at a certain moment and under certain conditions, taking into account his/her feelings about that moment. There are 20 questions in the trait anxiety scale. It is asked to measure an individual's trait anxiety. The trait anxiety scale includes questions about how the individual usually feels. The total score value obtained from each scale is between 20-80. A high score indicates a high level of anxiety and a low score indicates a low level of anxiety.
postoperative mobility | up to six months
  The effects of routine patient education and video-assisted mobilization training on postoperative mobility in patients undergoing coronary artery bypass graft surgery were investigated.
  Patient Mobility Scale and Observer Mobility were used to measure the level of postoperative mobility. The patient mobility and observer mobility scale consists of two parts: "Patient Mobility" and "Observer Mobility".
  The Patient Mobility Scale includes questions to measure the difficulty and pain experienced by the individual during activities such as turning from one side to the other in bed, sitting on the edge of the bed, standing up on the edge of the bed and walking in the patient room. It was evaluated using a 15 cm visual analog and verbal statements were included at the bottom.
  The Observer Mobility Scale consists of the assessment of 4 postoperative activities including turning, sitting, standing and walking. The patient's dependence or independence on the nurse is calculated.
postoperative pain | up to six months
  The effects of routine patient education and video-assisted mobilization training on postoperative mobility in patients undergoing coronary artery bypass graft surgery were investigated.
  Patient Mobility Scale and Observer Mobility were used to measure the level of postoperative mobility. The patient mobility and observer mobility scale consists of two parts: "Patient Mobility" and "Observer Mobility".
  The Patient Mobility Scale includes questions to measure the difficulty and pain experienced by the individual during activities such as turning from one side to the other in bed, sitting on the edge of the bed, standing up on the edge of the bed and walking in the patient room. It was evaluated using a 15 cm visual analog and verbal statements were included at the bottom.
  The Observer Mobility Scale consists of the assessment of 4 postoperative activities including turning, sitting, standing and walking. The patient's dependence or independence on the nurse is calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Tosun, Tekirdağ, Teki̇rdağ, Turkey (Türkiye)